CLINICAL TRIAL: NCT03317652
Title: Effect of Sodium Nitroprusside on Cerebral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Niels Damkjær Olesen, Principal investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-17017045
Record Dates: First submitted 2017-10-03; First posted 2017-10-23 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sodium nitroprusside and CO2 reactivity (Experimental): The subject rests in the supine position throughout the study that lasts for approximately three hours.
  Interventions are:
  * Hyperventilation
  * 6% CO2 breathing
  * Infusion of sodium nitroprusside
  Interventions: Other: Hyperventilation; Other: 6% CO2 breathing; Drug: Infusion of sodium nitroprusside

INTERVENTIONS:
Other: Hyperventilation — The subject is instructed to hyperventilate for 6 min to provoke a 0.7-1.2 kPa reduction in PaCO2, and the evaluation is repeated if the reduction in PaCO2 is not within this interval. The order of hyperventilation and 6% CO2 breathing is randomized.
  Other Names: Evaluation of CO2 reactivity, hyperventilation
Other: 6% CO2 breathing — The subject breathes a mixture of 6% CO2 (with 21% O2 and 73% N2) from a bag and a face mask for 6 minutes. The order of hyperventilation and 6% CO2 breathing is randomized.
  Other Names: Evaluation of CO2 reactivity, 6% CO2 breathing
Drug: Infusion of sodium nitroprusside — Using incremental intravenous infusion of sodium nitroprusside MAP is reduced by 20% (15%-25%) and then by 40% (35%-45%, MAP minimally at 50 mmHg).

SUMMARY:
The brain has a high energy demand and requires continuous blood flow. The blood flow to the brain appears to be unaffected by small changes in blood pressure, but brain blood flow may be reduced by a large reduction in blood pressure. Large reductions in blood pressure are common during anesthesia or bleeding. It is unclear, however, how a given reduction in blood pressure affects blood flow to the brain.

In this study, medicine called sodium nitroprusside is used to dilate blood vessels and reduce blood pressure in twenty healthy young men. The study will evaluate whether blood flow to the brain is affected when sodium nitroprusside is used to induce a moderate and a large reduction in blood pressure. Blood flow to the brain is evaluated using ultrasound on the neck.

During breathing, oxygen is inhaled and carbon dioxide is exhaled. Carbon dioxide increases brain blood flow whereby changes in respiration can affect the blood flow to the brain. Sodium nitroprusside causes mild hyperventilation, whereby more carbon dioxide is exhaled, which will contribute to a reduction in brain blood flow. Thus, the study will also evaluate how brain blood flow is affected by hyperventilation and by breathing a mix of air and carbon dioxide.

DETAILED DESCRIPTION:
Background Cerebral autoregulation is generally considered to maintain cerebral blood flow (CBF) if mean arterial pressure (MAP) is between 60 and 150 mmHg. Yet, it is controversial whether there is a plateau for CBF. Thus, blood velocity of the middle cerebral artery (MCA Vmean), as an index of CBF, is affected by pharmacological changes in MAP between approximately 40-125 mmHg. In contrast, internal carotid artery blood flow is unaffected by a moderate decrease in blood pressure.

The brain is supplied by the internal carotid and vertebral arteries that have different regulation with higher CO2 reactivity and larger orthostatic reduction for the internal carotid than the vertebral artery. The different regulation of the two arteries may reflect higher sympathetic innervation of arteries that originate from the internal carotid artery than those of the vertebral artery. The internal carotid artery may contribute to cerebral autoregulation as the vessel dilates during a moderate decrease in MAP while internal carotid artery blood flow is maintained. The arterial CO2 tension (PaCO2) is an important regulator of CBF and also maintenance of central blood volume and cardiac output is important for regulation of CBF. In the present study, internal carotid and vertebral artery blood flow is evaluated using duplex ultrasound in 20 healthy men when MAP is reduced by sodium nitroprusside, a potent short-lasting vasodilator.

Objective The purpose of the study is to evaluate whether CBF is affected by 20% and 40% reductions in MAP by sodium nitroprusside. The CO2 reactivity of the internal carotid and vertebral arteries is evaluated in order to control for hyperventilation during sodium nitroprusside induced hypotension. Further, the study will evaluate whether changes in internal carotid and vertebral artery blood flow by a 40% reduction in MAP are different and whether the arteries have different CO2 reactivity. Lastly, the study will evaluate whether the slope of the linear regression of CBF and MAP is higher for the evaluations when MAP is reduced by 40% and 20% than that of the evaluations at baseline and when MAP is reduced by 20%.

Hypotheses

* Sodium nitroprusside-induced reduction in MAP by 40% reduces CBF
* Sodium nitroprusside-induced reduction in MAP by 20% reduces CBF
* Sodium nitroprusside-induced reduction in MAP by 40% causes a larger relative reduction in internal carotid artery blood flow than that of the vertebral artery
* The CO2 reactivity of the internal carotid artery is higher than that of the vertebral artery
* The slope of linear regression of MAP and CBF at the evaluations when MAP is reduced by 20% and 40% by sodium nitroprusside is higher than that of the evaluations at baseline and when MAP is reduced by 20%

Methods The study will include 20 healthy men. The experiment lasts for approximately three hours and the subject must be fasting for at least 4 hours, have abstained from alcohol and caffeine for 12 hours and rigorous exercise for 24 hours. Before the start of the experiment, the internal carotid and vertebral arteries are evaluated and in case the vessels can not be visualized, e.g. because of high carotid bifurcation, the subject will not be able to participate in the study. The subject rests in the supine position throughout the study.

Measurements A catheter is placed in the radial or brachial artery on the non-dominant arm for evaluation of arterial pressure and gas variables. Total volume of blood sampled is less than 25 ml. A long line is placed in a cubital vein and advanced to the subclavian vein for infusion of sodium nitroprusside. The arterial pressure measurement is used for evaluation of stroke volume, cardiac output, and total peripheral resistance by modified pulse contour analysis. Heart rate is evaluated by electrocardiogram lead II. Forehead skin oxygenation and blood flow is evaluated close to the hairline using Laser Doppler flowmetry with an integrated oxygenation sensor at a depth of 1-2 mm in an area of approximately 9 mm^2. Cerebral and biceps muscle oxygenation are evaluated using near-infrared spectroscopy . Transcranial Doppler is used to evaluate MCA Vmean. At a constant diameter of the MCA, changes in blood velocity reflect those of regional CBF, but the diameter may be affected by changes in MAP and PaCO2.

Changes in central blood volume are evaluated by recording of thoracic electric admittance. Central hemodynamics, MCA Vmean, electrocardiogram, and skin oxygenation and blood flow is recorded at 100 hertz, cerebral and muscle oxygenation is recorded at 0.1 hertz, and thoracic admittance at 0.25 hertz and saved on a pc.

Internal carotid and vertebral artery blood flow is evaluated unilaterally on the neck using duplex ultrasound. Evaluation is in the longitudinal section 1-2 cm distal to the carotid bifurcation and the vertebral artery is evaluated between the transverse processes of C2-5 with the head turned approximately 30⁰ to the contralateral side. In order to limit the influence of ventilation, two recordings of approximately 20 s of both arteries are conducted at each level of MAP and the mean is reported. A frequency of 8-12 megahertz is used and gain is set as high as possible while vessel lumen is echo-free. Pulsed-wave Doppler at a stable angle ≤ 60º determined the angle-corrected time averaged maximum flow velocity (TAVMAX), that corresponds to twice the mean blood velocity. Diameter is assessed using automatic software to track the vessel wall and blood flow is: 0.125 * 60 * TAVMAX * π * diameter^2 and CBF is the sum of unilateral internal carotid and vertebral artery blood flow.

The CO2 reactivity of the internal carotid and vertebral artery is: change in blood flow *100 / change in PaCO2 * baseline blood flow using individual linear regression for the evaluations during normo-, hypo-, and hypercapnia. The CO2 reactivity of MCA Vmean and cerebral oxygenation is evaluated similarly and measurements during sodium nitroprusside infusion are corrected for changes in PaCO2 from baseline using the CO2 reactivity to hypocapnia.

Procedures Baseline evaluation at rest is conducted at least 30 min after placement of catheters. Subsequently, the CO2 reactivity is evaluated during hypo- and hypercapnia in random order. Hypocapnia is attained by hyperventilation for 6 min to provoke a 0.7-1.2 kilopascal (kPa) reduction in PaCO2, and the evaluation is repeated if the reduction in PaCO2 is not within this interval. Hypercapnia is achieved by breathing 6% CO2 for 6 min.

Thereafter, sodium nitroprusside is infused to reduce MAP by 20% (15%-25%) and 40% (35%-45% and minimally MAP 50 mmHg at a maximal infusion rate of 10 µg/(kg*min)). Sodium nitroprusside is a short-acting, potent vasodilator that activates guanylate cyclase directly or by production of nitric oxide, causing relaxation of smooth muscle cells in arteries and veins. The effect of sodium nitroprusside is attained within 2 min, and the half-life is 2 min whereby the effect is short lasting. Sodium nitroprusside has no direct effect on CBF. Infusion of sodium nitroprusside is by an electronic infusion pump, at 0.25 µg/(kg*min) for one minute and increased by 0.25 µg/(kg*min) each minute. The effect on MAP is evaluated each minute before the infusion speed is increased. When a level of MAP is reached, MAP is maintained for another minute where after measurements are conducted during 2-3 min. When evaluations have been done at both levels of MAP, the infusion speed is reduced gradually in order to avoid so-called "rebound hypertension". At this time the experiment is finished and catheters are removed.

Statistics Trial size: In a similar study, sodium nitroprusside-induced reduction in MAP by 43% decreased CBF by 15% after correction for the decrease in PaCO2. A power calculation indicates that at least 14 subjects are required to detect a 15% reduction in CBF with a standard deviation of 18% when MAP is reduced by 40% by sodium nitroprusside with a 5% significance level and a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Male
* Age 18-35 years

Exclusion Criteria:

* Alcohol intake ≥ 420 g / week
* Body mass index below 18 kg/m^2 and above 25 kg/m^2
* Smoking
* Beard on the neck
* Chronic cardiac, lung, liver, kidney or metabolic disease that require medication
* Vitamin B12 deficiency
* Anemia
* Leber's hereditary optic neuropathy
* Tobacco-alcohol amblyopia
* Stenosis that obstructs ≥ 16% of the internal carotid artery
* Intake of sildenafil or vardenafil for 24 hours and tadalafil for 48 timer prior to the experiment
* Intake of monoamine oxidase inhibitors
* Neurologic disease considered to affect cerebral blood flow, including epilepsy and multiple sclerosis

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Change in cerebral blood flow from baseline to when MAP (mean arterial pressure) is decreased by 40% by sodium nitroprusside | Values are recorded during 2-3 min at 2 time points; at baseline and when MAP is reduced by 40% by sodium nitroprusside (approximately 2 hours after the baseline evaluation)
  Sum of unilateral internal carotid and vertebral artery blood flow [ml/min] by duplex ultrasound corrected for changes in arterial CO2 tension (PaCO2) from baseline

SECONDARY OUTCOMES:
Change in cerebral blood flow from baseline to when MAP is decreased by 20% by sodium nitroprusside | Values are recorded during 2-3 min at 2 time points; at baseline and when MAP is reduced by 20% by sodium nitroprusside (approximately 2 hours after the baseline evaluation)
  Sum of unilateral internal carotid and vertebral artery blood flow [ml/min] by duplex ultrasound corrected for changes in PaCO2 from baseline
Relative reduction in internal carotid artery blood flow as compared to that of the vertebral artery from baseline to when MAP is reduced by 40% by sodium nitroprusside | Values are recorded during 2-3 min at 2 time points; at baseline and when MAP is reduced by 40% by sodium nitroprusside (approximately 2 hours after the baseline evaluation)
  Internal carotid and vertebral artery blood flow [ml/min] by duplex ultrasound corrected for changes in PaCO2 from baseline
The CO2 reactivity of the internal carotid as compared to the vertebral artery | Values are recorded during 2-3 min at 3 time points; at baseline, during hyperventilation for 6 min (approx 60 min after the baseline evaluation) and during 6% CO2 breathing for 6 min (approximately 60 min after the baseline evaluation)
  The CO2 reactivity of the internal carotid and vertebral arteries as evaluated during baseline, hyperventilation, and 6% CO2 breathing as: change in blood flow *100 / (change in PaCO2 * baseline blood flow). Internal carotid and vertebral artery blood flow [ml/min] by duplex ultrasound and PaCO2 [kilopascal] by arterial gas analysis
Comparison of the slope of linear regression of MAP and cerebral blood flow for the evaluations at baseline and when MAP is reduced by 20% by sodium nitroprusside and that of the evaluations when MAP is reduced by 20% and 40% | Values are recorded during 2-3 min at 3 time points; at baseline and when MAP is reduced by 20% and 40% by sodium nitroprusside (both approximately 2 hours after the baseline evaluation)
  Sum of unilateral internal carotid and vertebral artery blood flow [ml/min] by duplex ultrasound corrected for changes in PaCO2 from baseline and MAP [mmHg] by arterial cannulation

CONTACTS AND LOCATIONS:
Overall Officials: Niels D Olesen, MD, Principal Investigator — Department of Anesthesia, Rigshospitalet 2043, DK-2100 Copenhagen Ø, Denmark
Locations (1):
- Department of Anesthesia, Rigshospitalet 2043, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edvinsson L, Owman C. Sympathetic innervation and adrenergic receptors in intraparenchymal cerebral arterioles of baboon. Acta Neurol Scand Suppl. 1977;64:304-5. No abstract available. PMID 409067
- [Background] Evans DH. On the measurement of the mean velocity of blood flow over the cardiac cycle using Doppler ultrasound. Ultrasound Med Biol. 1985 Sep-Oct;11(5):735-41. doi: 10.1016/0301-5629(85)90107-3. PMID 2932831
- [Background] Henriksen L, Paulson OB. The effects of sodium nitroprusside on cerebral blood flow and cerebral venous blood gases. II. Observations in awake man during successive blood pressure reduction. Eur J Clin Invest. 1982 Oct;12(5):389-93. doi: 10.1111/j.1365-2362.1982.tb00685.x. PMID 6816609
- [Background] Hoiland RL, Ainslie PN. CrossTalk proposal: The middle cerebral artery diameter does change during alterations in arterial blood gases and blood pressure. J Physiol. 2016 Aug 1;594(15):4073-5. doi: 10.1113/JP271981. Epub 2016 Mar 24. No abstract available. PMID 27010010
- [Background] Jorgensen LG, Perko M, Perko G, Secher NH. Middle cerebral artery velocity during head-up tilt induced hypovolaemic shock in humans. Clin Physiol. 1993 Jul;13(4):323-36. doi: 10.1111/j.1475-097x.1993.tb00333.x. PMID 8370233
- [Background] LASSEN NA. Cerebral blood flow and oxygen consumption in man. Physiol Rev. 1959 Apr;39(2):183-238. doi: 10.1152/physrev.1959.39.2.183. No abstract available. PMID 13645234
- [Background] Lewis NC, Smith KJ, Bain AR, Wildfong KW, Numan T, Ainslie PN. Impact of transient hypotension on regional cerebral blood flow in humans. Clin Sci (Lond). 2015 Jul;129(2):169-78. doi: 10.1042/CS20140751. PMID 25697830
- [Background] Liu J, Zhu YS, Hill C, Armstrong K, Tarumi T, Hodics T, Hynan LS, Zhang R. Cerebral autoregulation of blood velocity and volumetric flow during steady-state changes in arterial pressure. Hypertension. 2013 Nov;62(5):973-9. doi: 10.1161/HYPERTENSIONAHA.113.01867. Epub 2013 Sep 16. PMID 24041946
- [Background] Lucas SJ, Tzeng YC, Galvin SD, Thomas KN, Ogoh S, Ainslie PN. Influence of changes in blood pressure on cerebral perfusion and oxygenation. Hypertension. 2010 Mar;55(3):698-705. doi: 10.1161/HYPERTENSIONAHA.109.146290. Epub 2010 Jan 18. PMID 20083726
- [Background] Meng L, Hou W, Chui J, Han R, Gelb AW. Cardiac Output and Cerebral Blood Flow: The Integrated Regulation of Brain Perfusion in Adult Humans. Anesthesiology. 2015 Nov;123(5):1198-208. doi: 10.1097/ALN.0000000000000872. PMID 26402848
- [Background] Panerai RB. Assessment of cerebral pressure autoregulation in humans--a review of measurement methods. Physiol Meas. 1998 Aug;19(3):305-38. doi: 10.1088/0967-3334/19/3/001. PMID 9735883
- [Background] Sato K, Fisher JP, Seifert T, Overgaard M, Secher NH, Ogoh S. Blood flow in internal carotid and vertebral arteries during orthostatic stress. Exp Physiol. 2012 Dec;97(12):1272-80. doi: 10.1113/expphysiol.2012.064774. Epub 2012 Jun 11. PMID 22689443
- [Background] Sato K, Sadamoto T, Hirasawa A, Oue A, Subudhi AW, Miyazawa T, Ogoh S. Differential blood flow responses to CO(2) in human internal and external carotid and vertebral arteries. J Physiol. 2012 Jul 15;590(14):3277-90. doi: 10.1113/jphysiol.2012.230425. Epub 2012 Apr 23. PMID 22526884
- [Background] Thomas KN, Lewis NC, Hill BG, Ainslie PN. Technical recommendations for the use of carotid duplex ultrasound for the assessment of extracranial blood flow. Am J Physiol Regul Integr Comp Physiol. 2015 Oct;309(7):R707-20. doi: 10.1152/ajpregu.00211.2015. Epub 2015 Jul 8. PMID 26157060
- [Background] Torella F, McCollum CN. Regional haemoglobin oxygen saturation during surgical haemorrhage. Minerva Med. 2004 Oct;95(5):461-7. PMID 15467521
- [Background] Verbree J, Bronzwaer AS, Ghariq E, Versluis MJ, Daemen MJ, van Buchem MA, Dahan A, van Lieshout JJ, van Osch MJ. Assessment of middle cerebral artery diameter during hypocapnia and hypercapnia in humans using ultra-high-field MRI. J Appl Physiol (1985). 2014 Nov 15;117(10):1084-9. doi: 10.1152/japplphysiol.00651.2014. Epub 2014 Sep 4. PMID 25190741
- [Background] Aaslid R, Markwalder TM, Nornes H. Noninvasive transcranial Doppler ultrasound recording of flow velocity in basal cerebral arteries. J Neurosurg. 1982 Dec;57(6):769-74. doi: 10.3171/jns.1982.57.6.0769. PMID 7143059

DOCUMENTS (2):
  • Study Protocol (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT03317652/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT03317652/SAP_001.pdf